CLINICAL TRIAL: NCT06513234
Title: Orelabrutinib Combined With Obinutuzumab as First-line Treatment for Marginal Zone Lymphoma：a Prospective Single Arm Trial
Brief Title: Combination of Orelabrutinib and Obinutuzumab in Untreated Marginal Zone Lymphomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024013
Record Dates: First submitted 2024-07-01; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-06

CONDITIONS: Marginal Zone Lymphoma
Keywords: Marginal Zone Lymphomas; orelabrutinib; obinutuzumab
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OG (Experimental): 6 cycles of OG regimen. Patients with CR/PR after 6 cycles of OG treatment will be treated with 18 cycles of single-agent orelabrutinib regimen. Orelabrutinib 150mg QD
  Interventions: Drug: Orelabrutinib and obinutuzumab

INTERVENTIONS:
Drug: Orelabrutinib and obinutuzumab — Orelabrutinib and obinutuzumab 6cycles ;orelabrutinib 150mg

SUMMARY:
This is a prospective single arm phase II study, and the purpose of this study is to evaluate the safety and efficacy of orelabrutinib combined with obinutuzumab a in untreated marginal zone lymphoma. It is planned to recruit 45 patients. The primary endpoint is the complete remission rate at 12 months.

DETAILED DESCRIPTION:
Marginal zone lymphomas (MZL) are a type of lymphoma that originates from the marginal zone tissue of the lymphoid follicles (Mucosa-associated lymphoid tissue, MALT), and include three subtypes: MALT lymphoma, nodal MZL, and splenic MZL. For patients with marginal zone lymphoma who have indications for systemic anti-tumor treatment, therapeutic options include rituximab monotherapy or more intensive immunochemotherapy regimens in combination with bendamustine, chlorambucil, CHOP regimen (cyclophosphamide, vincristine, doxorubicin, prednisone), etc.

This is a prospective, phase II, single-arm clinical study to initially explore the efficacy and safety of Orelabrutinib combined with obinutuzumab in patients with previously untreated marginal zone lymphoma. The patients will be treated with 6 cycles of OG regimen. Patients with CR/PR after 6 cycles of OG treatment will be treated with 18 cycles of single-agent orelabrutinib regimen.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥18 years, gender unrestricted;

  * Histopathologically confirmed CD20-positive marginal zone lymphoma including MALT, SMZL, NMZL;
  * MZL that has progressed, recurred, or is unsuitable for local treatment after previous local therapy (local treatments include surgery, radiotherapy, Helicobacter pylori treatment, hepatitis C treatment);
  * ECOG performance status score of 0-2.
  * Major organ functions meet the following criteria: a) Complete blood count: Absolute neutrophil count ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥75g/L; if accompanied by bone marrow involvement, absolute neutrophil count ≥1.0×10^9/L, platelets ≥50×10^9/L, hemoglobin ≥50g/L; b) Blood biochemistry: Total bilirubin ≤1.5 times the upper limit of normal (ULN), AST or ALT ≤2 times ULN; serum creatinine ≤1.5 times ULN; serum amylase ≤ULN; c) Coagulation function: International normalized ratio (INR) ≤1.5 times ULN.
  * Life expectancy ≥3 months;
  * Voluntarily sign a written informed consent form before the trial screening.

Exclusion Criteria:

* Currently or previously having other malignant tumors, unless radical treatment has been performed and there is evidence of no recurrence or metastasis within the last 5 years;
* Lymphoma involving the central nervous system or transforming into a higher grade;
* Having uncontrollable or significant cardiovascular diseases, including: a) New York Heart Association (NYHA) class II or above congestive heart failure, unstable angina, myocardial infarction within 6 months before the first administration of the study drug, or arrhythmias requiring treatment at the time of screening, with a left ventricular ejection fraction (LVEF) <50%; b) Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, unclassified cardiomyopathy); c) A history of clinically significant QTc interval prolongation, or a QTc interval >470ms in females and >450ms in males during the screening period; d) Subjects with symptomatic or medication-requiring coronary artery heart disease; e) Subjects with difficult-to-control hypertension (despite lifestyle improvements and the use of reasonable, tolerable, and adequate doses of one or three or more antihypertensive drugs [including diuretics] for more than 1 month, blood pressure is still not at the standard, or it is only effectively controlled when taking four or more antihypertensive drugs).
* Active bleeding within 2 months before screening, or currently taking anticoagulant drugs, or the investigator believes there is a definite bleeding tendency;
* Active infection or uncontrolled HBV (positive for HBsAg and/or HBcAb with positive HBV DNA titer), positive for HCV Ab, HIV/AIDS, or other serious infectious diseases.
* Any other conditions deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-11 (Estimated); Primary Completion 2026-06-21 (Estimated); Study Completion 2029-06-21 (Estimated)

PRIMARY OUTCOMES:
the complete response rate | At 12 months.
  CRR is defined as the proportion of patients with a response of CR

SECONDARY OUTCOMES:
CRR | At the end of induction therapy(6cycles). 28days/cycle
  CRR is defined as the proportion of patients with a best response of CR
ORR | At 12 months.
  The ORR is defined as the proportion of patients with a response of CR
BOR | At 12 months.
  The BOR is defined as the proportion of patients with a best response of CR or PR
2 years progression-free survival | From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
2 years overall survival | From date of signing the informed consent until the date of death from any cause, whichever came first, assessed up to 2 years]
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
TTR | Up to 2 years
  TTR is defined as the time from registration to the first response.
Duration of Response (DOR) | Up to 2 years
  Duration of response as defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
The occurrence of adverse events and serious adverse events | One month after discontinuation of treatment
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.

CONTACTS AND LOCATIONS:
Locations (1):
- China Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, China